CLINICAL TRIAL: NCT06317493
Title: Using Pupillometry to Assess Hearing Thresholds in Young Children With Hearing Impairment
Brief Title: Hearing Impairment in Children: Pupillometry and Hearing Thresholds Assessment
Status: Recruiting | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 15/2021
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Hearing Impaired Children
Keywords: Pupillometry; Hearing threshold; Pediatric cochlear implants
MeSH Terms: interventions — Stimuli Responsive Polymers

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Hearing threshold without aids: Case group with hearing impairment (HI) (hearing threshold >35 dB) without aids
  Interventions: Other: Stimuli
- Hearing threshold with cochlear implant: Case group with hearing threshold corrected with cochlear implant (CI)
  Interventions: Other: Stimuli
- Hearing threshold with aids: Case group with hearing threshold corrected with hearing aids
  Interventions: Other: Stimuli
- Control group: Control group of normally hearing age-matched children
  Interventions: Other: Stimuli

INTERVENTIONS:
Other: Stimuli — Auditory Stimuli: Pure tone bursts with main frequencies of 500, 1000, 2000, and 4000 Hz. Each tone will be presented at 10dB above the estimated individual threshold per frequency and compared to the responses to trials without auditory stimuli. Auditory stimulus duration: 25ms, there is 200ms baseline period before each trial, and 2000 ms interstimulus interval.
  Visual stimuli: an animated movie adapted for the age and controlled for luminosity levels.
  Pupil data will be collected through a "Tobii PRO" screen-based eye-tracker that measures eye-movements and pupil dilation using the infrared light cameras.

SUMMARY:
The results of the previous study on auditory effort in young children with cochlear implants show that pupils respond to the presence or the absence of the perceived stimuli. The investigators hypothesize that the perceived sounds will elicit increased pupil dilation compared to the non-perceived sounds and that the hearing threshold as measured with pure tone audiometry will correlate to the results in pupillometry test. The investigators hypothesize that the effect will be visible in all testing groups albeit the relative increase of pupil size with age. Hypothesis confirmed, the investigators will develop a standardised procedure for the auditory signal detection using pupillometry. Such a procedure could represent an important bridge between automatic and behavioral hearing tests. With a more precise test of auditory threshold of young children, post-operative monitoring and fitting of cochlear implants or hearing aids, and rehabilitation procedures, could be considerably more targeted and consequentially more efficient.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected-to-normal vision
* No history of relevant neurological or psychiatric concomitant disease
* Age: 4-36 months
* At least 1 months of more after initial fitting of the CI or hearing aid (only for aided subjects)

Exclusion Criteria:

* Developmental disorders
* Unwillingness of the subject to participate further

Ages: 4 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants with and without hearing impairment
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-01-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity index of pupillometry test | Within 30 minutes from enrolment
  The peak and the average pupil dilation will be defined for each trial and the difference between trials below and above the threshold will be defined within each block. The difference between the trials with and without audible stimuli will be assessed using the multiple corrected t- tests. The sensitivity index of the pupillometric exam compared to the audiometry results will be computed for the whole group using a signal detection analysis.

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (4):
  - UOC Otorinolaringoiatria, Padua
  - Università degli Studi di Perugia, Perugia
  - Ospedale Martini, Torino
  - Institute for Maternal and Child Health - IRCCS "Burlo Garofolo", Trieste
- Univeristy Medical Center, Ljubljana, Slovenia